CLINICAL TRIAL: NCT04390620
Title: Assessment of DAFILON® Suture Material in Oral Surgery (Mucosal Sutures). A Prospective, Single Arm Observational Study in Daily Practice
Brief Title: Assessment of DAFILON® Suture Material in Oral Surgery (Mucosal Sutures)
Acronym: MUCODA
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1912
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Oral Surgery; Tooth Extraction; Dental Implants
Keywords: oral surgery; mucosal closure; complication rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MUCODA: DAFILON - sterile, monofilament, non-absorbable surgical suture material produced from Polyamide
  Interventions: Device: Mucosal Closure

INTERVENTIONS:
Device: Mucosal Closure — mucosal closure in oral surgery (mucosal sutures)

SUMMARY:
In this non-interventional study (NIS) a polyamide non-absorbable suture (Dafilon) will be evaluated for oral surgery (mucosal closure after e.g. wisdom teeth extraction, implant surgery, etc.) in adult patients

DETAILED DESCRIPTION:
In this non-interventional study (NIS) a polyamide non-absorbable suture (Dafilon) will be evaluated for oral surgery (mucosal closure after e.g. wisdom teeth extraction, implant surgery, etc.) in adult patients.

The aim of this NIS is to collect systematically and proactively different clinical parameters regarding safety, effectiveness and performance of Dafilon suture material under the daily routine clinical practice when is intended to be used for oral surgery. All patients enrolled will be prospectively followed until suture removal, which takes place 10 ± 5 days post-operatively (and post-operatively depending on routine clinical practice of each hospital).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing mucosal wound closure using Dafilon as suture material in oral surgery (in the event that more than one incision is performed in the same patient, only one incision will be included).
* Written informed consent regarding the data collection for the PMCF.

Exclusion Criteria:

* Emergency surgery.
* Oral surgery procedures requiring bone regeneration.
* Pregnancy.
* Patients taking medication that might affect wound healing.
* Patients with hypersensitivity or allergy to the suture material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
incidence of combined postoperative complications Grade I and Grade II | 10 ± 5 days postoperatively (suture removal)
  combined incidence of postoperative complications Grade I & II on a Five Point scale defined by Askar et al. (Grade I: postoperative dentinal hypersensitivity / Oral candidiasis / Angular cheilitis / Exaggerated swelling defined as postoperative enlargement of tissues that exceeds the normal limits associated with a given surgical procedure / Delayed wound healing defined as an unusual deviation from the normal course of healing / Mild postoperative bleeding defined as the presence of small amount of blood in the oral cavity, usually mixed with saliva; Grade II: Flap dehiscence / Membrane exposure / Localized infection of the surgical site / Graft necrosis)

SECONDARY OUTCOMES:
Incidence of individual postoperative complications | until suture removal 10 ± 5 days postoperative
  incidence of postoperative complications of Grade I - V on a Five Point scale defined by Askar et al. (Grade I & II see Primary Outcome; Grade III: Fever / Skin rash / Neuropraxia/paresthesia / Trimus / Osteomyelitis / Septicemia / Sinusitis / Alveolar osteitis / Chymosis / Excessive and severe bleeding / Prolonged exaggerated swelling; Grade IV: Major complications that required immediate hospitalization such as drug induced anaphylaxis or septicemia; Grade V: Major complications that led to irreversible damage such neurotmesis and axonotmesis)
Pain assessment using the visual analogue scale (VAS 1-100) | at suture removal 10 ± 5 days postoperative
  This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain".
Satisfaction of the patient using the visual analogue scale (VAS 1-100) | at suture removal 10 ± 5 days postoperative
  This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "completely satisfied" and "100" at the opposite end representing "not at all satisfied".
Wound healing assessment using the visual analogue scale (VAS 1-100) | at suture removal 10 ± 5 days postoperative
  This parameter will be noted by the surgeon using the Visual Analogue Scale (VAS) which state "0" at one end representing "very good wound healing" and "100" at the opposite end representing "very bad wound healing".
knot security | intraoperative
  Evaluation of Knot security with the 5 evaluation levels 'excellent', 'very good', 'good', 'satisfied' and 'poor' into the evaluation scores 5, 4, 3, 2 and 1,
tensile strength | intraoperative
  Evaluation of tensile strength with the 5 evaluation levels 'excellent', 'very good', 'good', 'satisfied' and 'poor' into the evaluation scores 5, 4, 3, 2 and 1,
knot run down | intraoperative
  Evaluation of knot run down with the 5 evaluation levels 'excellent', 'very good', 'good', 'satisfied' and 'poor' into the evaluation scores 5, 4, 3, 2 and 1,
tissue drag | intraoperative
  Evaluation of tissue drag with the 5 evaluation levels 'excellent', 'very good', 'good', 'satisfied' and 'poor' into the evaluation scores 5, 4, 3, 2 and 1,
pliability | intraoperative
  Evaluation of pliability with the 5 evaluation levels 'excellent', 'very good', 'good', 'satisfied' and 'poor' into the evaluation scores 5, 4, 3, 2 and 1,

OTHER OUTCOMES:
Bacterial contamination of the thread | at suture removal 10 ± 5 days postoperative
  optional
Pain assessment using the visual analogue scale (VAS 1-100) | at follow-up up to five months postoperative
  Optional: This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain".
Satisfaction of the patient using the visual analogue scale (VAS 1-100) | at follow-up up to five months postoperative
  Optional: This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "completely satisfied" and "100" at the opposite end representing "not at all satisfied".
Wound healing assessment using the visual analogue scale (VAS 1-100) | at follow-up up to five months postoperative
  Optional: This parameter will be noted by the surgeon using the Visual Analogue Scale (VAS) which state "0" at one end representing "very good wound healing" and "100" at the opposite end representing "very bad wound healing".
Cosmetic outcome assessed by the physician using the visual analogue scale (VAS 1-100) | at follow-up up to five months postoperative
  Optional: This parameter will be noted by the surgeon using the Visual Analogue Scale (VAS) which state "0" at one end representing "very good cosmetic outcome" and "100" at the opposite end representing "very bad cosmetic outcome".

CONTACTS AND LOCATIONS:
Overall Officials: Nils Weyer, Dr. med., Principal Investigator — Praxisklinik für Mund-, Kiefer- und Gesichtschirurgie Ästhetische und Plastische Chirurgie
Locations (2):
- Praxisklinik für Mund-, Kiefer- und Gesichtschirurgie, Ästhetische und Plastische Chirurgie, Esslingen am Neckar, Germany
- Universitat Internacional de Catalunya (UIC), Barcelona, Spain